CLINICAL TRIAL: NCT03590392
Title: A Phase I Study to Determine the Safety and Immunogenicity of the Candidate Chikungunya Virus (CHIKV) Vaccine ChAdOx1 Chik in Healthy Adult Volunteers
Brief Title: Safety and Immunogenicity of a Candidate CHIKV Vaccine (CHIK001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHIK001
Record Dates: First submitted 2018-06-05; First posted 2018-07-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-07

CONDITIONS: Chikungunya Fever
Keywords: Vaccine; Chikungunya Virus; Chikungunya Fever
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1 volunteers (n= 6) will be administered ChAdOx1 Chik, 5 x 10^9 vp through intramuscular route.
  Interventions: Biological: ChAdOx1 Chik
- Group 2 (Experimental): Group 2 volunteers (n= 9) will be administered ChAdOx1 Chik, 2.5 x 10^10 vp through intramuscular route.
  Interventions: Biological: ChAdOx1 Chik
- Group 3 (Experimental): Group 3 volunteers (n= 9) will be administered ChAdOx1 Chik, 5 x 10^10 vp through intramuscular route.
  Interventions: Biological: ChAdOx1 Chik

INTERVENTIONS:
Biological: ChAdOx1 Chik — ChAdOx1 Chik, a replication-deficient simian adenoviral vector expressing CHIKV antigens.

SUMMARY:
A phase I dose escalation study to assess the safety and immunogenicity of the candidate vaccine ChAdOx1 Chik in healthy volunteers.

Volunteers will be recruited and vaccinated in Oxford, England.

All vaccinations will be administered intramuscularly. Three different doses will be tested (5x10^9 vp, 2.5x10^10 vp and 5x10^10vp).

The total duration of the study will be 26 weeks from the day of enrolment for all volunteers.

DETAILED DESCRIPTION:
This is a phase I, open label, dose escalation trial to assess the safety and immunogenicity of the ChAdOx1 Chik vaccine in healthy volunteers

There will be 3 study groups with a total of 24 volunteers. ChAdOx1 Chik will be administered intramuscularly as a single vaccination at 3 different doses: 5x10^9 vp (group 1), 2.5x10^10 (group 2) and 5x10^10 vp (group 3)

Vaccination of groups will be sequential from Group 1 to Group 3 with interim safety reviews prior to dose escalation

Volunteers will be recruited and undergo screening, vaccination and follow-up visits at the trial site. Blood samples for safety and immunology purposes will be performed on the visit time points indicated in the schedule of attendances.

Safety will be assessed by the frequency, incidence and nature of adverse events and serious adverse events arising during the study.

Immune responses will be assessed pre and post vaccination procedure at different time points throughout the trial

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 to 50 years
2. Able and willing (in the Investigator's opinion) to comply with all study requirements
3. Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
4. For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination
5. Agreement to refrain from blood donation during the course of the study
6. Provide written informed consent

Exclusion Criteria:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
2. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccine).
3. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
4. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
5. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
6. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
7. Any history of anaphylaxis in relation to vaccination
8. Pregnancy, lactation or willingness/intention to become pregnant during the study
9. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
10. History of serious psychiatric condition likely to affect participation in the study
11. Bleeding disorder (eg. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
12. Any other serious chronic illness requiring hospital specialist supervision
13. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
14. Suspected or known injecting drug abuse in the 5 years preceding enrolment
15. Seropositive for hepatitis B surface antigen (HBsAg)
16. Seropositive for hepatitis C virus (antibodies to HCV)
17. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
18. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
19. Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate
20. Prior exposure to CHIKV (serology will be requested at the discretion of the investigator)
21. Travel to a CHIKV endemic region throughout the duration of the participants enrolment in the Study and within the preceding 30 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited and unsolicited local and systemic adverse events | Solicited and Unsolicited AEs will be collected for 28 days. SAEs will be collected from enrolment until the end of the follow-up period (i.e 6 months)
  Occurrence of solicited and unsolicited local and systemic adverse events

SECONDARY OUTCOMES:
Measures of immunogenicity to the ChAdOx1 Chik in healthy adults volunteers | Up to 26 weeks
  Measures of immunogenicity to the ChAdOx1 Chik in healthy adults volunteers. Immunogenicity will be assessed by ELISA and ELISpot assays on the following days: 0 (vaccination visit), 14, 28, 56, and 182.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V Hill, DPhill FRCP, Principal Investigator — Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Folegatti PM, Harrison K, Preciado-Llanes L, Lopez FR, Bittaye M, Kim YC, Flaxman A, Bellamy D, Makinson R, Sheridan J, Azar SR, Campos RK, Tilley M, Tran N, Jenkin D, Poulton I, Lawrie A, Roberts R, Berrie E, Rossi SL, Hill A, Ewer KJ, Reyes-Sandoval A. A single dose of ChAdOx1 Chik vaccine induces neutralizing antibodies against four chikungunya virus lineages in a phase 1 clinical trial. Nat Commun. 2021 Jul 30;12(1):4636. doi: 10.1038/s41467-021-24906-y. PMID 34330906